CLINICAL TRIAL: NCT03326037
Title: Study of The Association of Mutations in The NPHS2 Gene and Nephrotic Syndrome in Children and Adults in Middle East
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: AHMED ABDULQADER HAMMOUDA ABOU SHALL (Other)
Collaborators: Kuwait University (Other); Assiut University (Other)
Responsible Party: Sponsor-Investigator, AHMED ABDULQADER HAMMOUDA ABOU SHALL, Senior nephrology registrar, Assiut University
Organization: Assiut University (Other)
Other Study IDs: MG03/15
Record Dates: First submitted 2017-10-22; First posted 2017-10-30 (Actual); Last update posted 2019-01-10 (Actual); Status verified 2019-01

CONDITIONS: Nephrotic Syndrome
Keywords: Nephrotic Syndrome; NPHS2 gene mutation; disease association
MeSH Terms: conditions — Nephrotic Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — Saliva and blood sampling and DNA extraction
  After obtaining informed consent from parents of children and adults, 3 ml of blood will be collected from children and in the event that the patients or their parents refuse then buccal swabs will be collected from children, and 5ml of blood will be collected from adults. The buccal swabs will be processed to extract DNA and stored at -20 till time of genetic analysis. Peripheral blood samples will be collected in EDTA anticoagulated tubes and DNA will be extracted according to standard methods using QIAGEN DNA blood mini kit (QIAGEN) and stored at 20 till time of analysis.
  Genotyping Genotyping of the NPHS2 variant rs61747728 will be performed by Real-time TaqMan Allelic Discrimination Assay (Life technologies, CA, USA) according to standard manufacturer protocols. Allelic discrimination analysis will be performed and analyzed using ABI 7500 Fast Real-time PCR system SDS software (Life technologies, CA, USA)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Genetic: Genotyping of the NPHS2 variant rs61747728 — Genotyping of the NPHS2 variant rs61747728 will be performed by Real-time TaqMan Allelic Discrimination Assay (Life technologies, CA, USA) according to standard manufacturer protocols. Allelic discrimination analysis will be performed and analyzed using ABI 7500 Fast Real-time PCR system SDS software (Life technologies, CA, USA)

SUMMARY:
Nephrotic syndrome (NS) represents one of the most common diagnoses in pediatric and adult nephrology, with a prevalence of 16 per 100,000 children and 3 per 100,000 adults in Western countries.

In most cases, the pathogenesis of NS remains elusive, and the clinical phenotype of patients does not allow discrimination among different causes. Thus, children with NS are usually treated with corticosteroids before a biopsy is taken, and approximately 80% of them respond to such a treatment. According to this observation, pediatric NS has been separated into two broad categories; Steroid-Sensitive Nephrotic Syndrome (SSNS) and Steroid-Resistant Nephrotic Syndrome (SRNS). In both these categories the biopsy result is usually Minimal Change Disease (MCD) while a few may show Focal and Segmental Glomerulosclerosis (FSGS). Although children affected by SSNS have good long-term prognosis, most patients with SRNS progress to End Stage Renal Disease (ESRD) within 2-10 years of diagnosis .

In adults a biopsy diagnosis of FSGS is more common than in children and more patients will not respond to corticosteroids alone and will need additional immunosuppressant medication. About 40% will progress to ESRD within 10 years .

Currently, at least 19 genes have been clearly identified with association to SRNS harboring ~300 independent mutations, conferring a considerable genetic heterogeneity to the disorder.

Genetic testing is emerging as a useful diagnostic tool in SRNS as it has implications for clinical course, treatment response, risk for posttransplant proteinuria and prenatal diagnosis. An approach for genetic testing based on the current evidence seems cost-effective and may help in the best possible management of SRNS .

The NPHS2 gene, is located on chromosome 1 and is also known as the Podocin gene. It encodes the podocin protein. Podocin is a 383-amino acid lipid-raft-associated protein localized at the slit diaphragm, where it is required for the structural organization and regulation of the glomerular filtration barrier. Its interaction with other slit diaphragm proteins eg. nephrin, NEPH1, CD2AP and TRPC6 is important in mechanosensation signaling, podocyte survival, cell polarity, and cytoskeletal organization .

.

It has been reported that variants in the NPHS2 gene are associated with NS .

The commonly studied rs61747728 NPHS2 gene polymorphism also known as p.R229Q has been reported to be associated with NS and SRNS .

However others have failed to report an association , which might be due to population differences.

The rs61747728 is a non-synonymous variant found on exon 5 which is suggested to be involved in in altering the functional properties of podocin in vitro and possibly in vivo .

The investigators will therefore investigate the frequency of the p.R229Q variant in Middle East patients with NS.

Genetic analysis will have important implications in several aspects:-

1. Understanding the biology of the disease in this part of the world.
2. Counselling patients about their clinical course and what medication they will respond to.
3. Counselling patients about the possibility of a kidney transplant sooner in their disease course

DETAILED DESCRIPTION:
Aim of the work:

The aim of this study is:

1. To identify any relationship between NPHS2 gene mutations and NS in children and adults in Middle East.
2. To study the relationship of mutations in this gene with the clinical presentation, clinical coarse and response to treatment in these patients and compare it with patients without mutations in this gene.
3. To compare our results with similar data from other World populations/ethnic groups.
4. To share our results with the treating clinicians so that counselling of the patients can be done in terms of treatment, prognosis and family screening.

Anticipated outcome and benefit :

With the increasing number of patients with NS in Middle East and the higher number of consanguineous marriages as compared to other societies, the investigators are sure that many gene mutations will be uncovered that may be the same as the previously reported genes or new novel genes.

In either case the investigators would have studied the genetic predisposition in our patient population and helped the nephrologists in taking appropriate treatment decisions.

The investigators expect a total of 150 patients with NS in both children and adults. About 20% will be from the pediatric population with MCD, while about 80% will be adults with predominantly FSGS.

Patient Recruitment:

This study will include patients referred to the nephrology departments in the major hospitals in Kuwait- Mubarak,Amiri,Farwaniya, Adan and Jahra Hospitals. Both children and adults of all ages.

This study will also include patients referred to the nephrology departments in Assuit university hospitals and all Upper Egypt hospitals Both children and adults of all ages,

Procedures:

Saliva and blood sampling and DNA extraction

After obtaining informed consent from parents of children and adults, 3 ml of blood will be collected from children and in the event that the patients or their parents refuse then buccal swabs will be collected from children, and 5 ml of blood will be collected from adults.All patients will be fully informed about the methods of blood sampling or buccal swabs and A written consent will be obtained from adult patients and parents of childrens. The buccal swabs will be processed to extract DNA and stored at -20 till time of genetic analysis. Peripheral blood samples will be collected in EDTA anticoagulated tubes and DNA will be extracted according to standard methods using QIAGEN DNA blood mini kit (QIAGEN) and stored at 20 till time of analysis.

Genotyping :

Genotyping of the NPHS2 variant rs61747728 will be performed by Real-time TaqMan Allelic Discrimination Assay (Life technologies, CA, USA) according to standard manufacturer protocols. Allelic discrimination analysis will be performed and analyzed using ABI 7500 Fast Real-time PCR system SDS software (Life technologies, CA, USA).

Statistical analysis

Basic statistical analysis will performed using SPSS software (version 22; SPSS Inc, Chicago, IL, USA). The genetic analysis will be performed using the SNPassoc package from R software.

ELIGIBILITY:
Inclusion Criteria:

* Inclusions criteria in children:

All children who presented with acute onset of heavy proteinuria (>3 g/24hrs).

If a biopsy was performed then only a diagnosis of MCD or FSGS will be included after performing light microscopy, immunofluorescence or immunoperoxidase testing and electron microscopy. These studies will be reviewed by the primary investigator.

If a biopsy is not performed as is the case with many children, then the clinical and serological parameters should be consistent with MCD or FSGS as evidenced by the negativity of autoimmune and infectious markers.. The cut off age used in referring patients to adult nephrologists is 16 years.

Inclusions criteria in adults :

All patients with proteinuria of acute or gradual onset but has to be more than 1g/24hrs. A biopsy must have been performed and reviewed by the primary investigator and the results should be MCD/FSGS after applying all the aforementioned pathological studies.

Exclusion Criteria:

* 1) All patients diagnosed as MCD secondary to:-

  1. Drugs:NSAIDs (most common), antimicrobials, lithium, bisphosphonates, and penicillamine (many others).
  2. Cancer:haematological malignancies (most common), solid organ malignancies (rarely associated with MCD).
  3. Infections:(rarely):esp.TB,syphilis,HIV, HCV, mycoplasma.
  4. Atopy:30% of MCD patients.
  5. Immunizations.

     2) All patients diagnosed as FSGS secondary to:-

  <!-- -->

  1. Infection (podocyte invasion): HIV-associated nephropathy (HIVAN) , Parvovirus B19.
  2. Drugs (podocyte toxicity): Pmidronate, lithium, interferon, and heroin.
  3. Congenital or acquired nephron mass reduction: Renal dyplasia, reflux nephropathy, renovascular disease, partial or unilateral nephrectomy.
  4. Hyperfiltration as part of disease process: Morbid obesity, diabetic nephropathy, pre-eclampsia, sickle cell disease.
  5. Any cause of glomerular disease with progressive scarring: Eg. Membranous GN, IgAN, Alport syndrome, thrombotic microangiopathy, vasculitis.

Ages: 2 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: This study will include patients referred to the nephrology departments in the major hospitals in Kuwait- Mubarak,Amiri,Farwaniya, Adan and Jahra Hospitals. Both children and adults of all ages.
  This study will also include patients referred to the nephrology departments in Assuit university hospitals and all Upper Egypt hospitals Both children and adults of all ages
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2016-10 (Actual); Primary Completion 2019-10 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Number of participants achieving NPHS2 gene mutations (frequency of p.R229Q polymorphic site) in patients with steroid-resistant nephrotic syndrome in comparison with steroid - sensitive nephrotic syndrome | Baseline to 2 years
  participants will be monitored for up to 2 years and classified as steroid -sensitive nephrotic syndrome or steroid - resistant nephrotic syndrome according to clinical response to steroid therapy ( 1 mg prednisolone /kg) for total 6 weeks.
  Renal biopsy will be done for all patients above 5 years of age (MCD and FSGS) were included.
  Blood sample or buccal swab will be collected from all patients and genotyping of the NPHS2 gene variant will be performed to report number of participants with NPHS2 gene mutations to share our results with the treating clinicians so that counselling of the patients can be done in terms of advising for kidney transplant sooner in their clinical course, prognosis and family screening.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine-Pathology Department, Hawalli, Kuwait

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] McKenzie LM, Hendrickson SL, Briggs WA, Dart RA, Korbet SM, Mokrzycki MH, Kimmel PL, Ahuja TS, Berns JS, Simon EE, Smith MC, Trachtman H, Michel DM, Schelling JR, Cho M, Zhou YC, Binns-Roemer E, Kirk GD, Kopp JB, Winkler CA. NPHS2 variation in sporadic focal segmental glomerulosclerosis. J Am Soc Nephrol. 2007 Nov;18(11):2987-95. doi: 10.1681/ASN.2007030319. Epub 2007 Oct 17. PMID 17942957
- [Result] Pollak MR. Inherited podocytopathies: FSGS and nephrotic syndrome from a genetic viewpoint. J Am Soc Nephrol. 2002 Dec;13(12):3016-23. doi: 10.1097/01.asn.0000039569.34360.5e. No abstract available. PMID 12444222
- [Result] Buscher AK, Weber S. Educational paper: the podocytopathies. Eur J Pediatr. 2012 Aug;171(8):1151-60. doi: 10.1007/s00431-011-1668-2. Epub 2012 Jan 13. PMID 22237399
- [Result] McCarthy HJ, Bierzynska A, Wherlock M, Ognjanovic M, Kerecuk L, Hegde S, Feather S, Gilbert RD, Krischock L, Jones C, Sinha MD, Webb NJ, Christian M, Williams MM, Marks S, Koziell A, Welsh GI, Saleem MA; RADAR the UK SRNS Study Group. Simultaneous sequencing of 24 genes associated with steroid-resistant nephrotic syndrome. Clin J Am Soc Nephrol. 2013 Apr;8(4):637-48. doi: 10.2215/CJN.07200712. Epub 2013 Jan 24. PMID 23349334
- [Result] Franceschini N, North KE, Kopp JB, McKenzie L, Winkler C. NPHS2 gene, nephrotic syndrome and focal segmental glomerulosclerosis: a HuGE review. Genet Med. 2006 Feb;8(2):63-75. doi: 10.1097/01.gim.0000200947.09626.1c. PMID 16481888
- [Result] Dusel JA, Burdon KP, Hicks PJ, Hawkins GA, Bowden DW, Freedman BI. Identification of podocin (NPHS2) gene mutations in African Americans with nondiabetic end-stage renal disease. Kidney Int. 2005 Jul;68(1):256-62. doi: 10.1111/j.1523-1755.2005.00400.x. PMID 15954915
- [Result] Zhang SY, Marlier A, Gribouval O, Gilbert T, Heidet L, Antignac C, Gubler MC. In vivo expression of podocyte slit diaphragm-associated proteins in nephrotic patients with NPHS2 mutation. Kidney Int. 2004 Sep;66(3):945-54. doi: 10.1111/j.1523-1755.2004.00840.x. PMID 15327385
- [Result] Rood IM, Deegens JK, Wetzels JF. Genetic causes of focal segmental glomerulosclerosis: implications for clinical practice. Nephrol Dial Transplant. 2012 Mar;27(3):882-90. doi: 10.1093/ndt/gfr771. Epub 2012 Feb 14. PMID 22334613
- [Result] Jain V, Feehally J, Jones G, Robertson L, Nair D, Vasudevan P. Steroid-resistant nephrotic syndrome with mutations in NPHS2 (podocin): report from a three-generation family. Clin Kidney J. 2014 Jun;7(3):303-5. doi: 10.1093/ckj/sfu028. Epub 2014 Apr 2. PMID 25852895
- [Result] Reiterova J, Safrankova H, Obeidova L, Stekrova J, Maixnerova D, Merta M, Tesar V. Mutational analysis of the NPHS2 gene in Czech patients with idiopathic nephrotic syndrome. Folia Biol (Praha). 2012;58(2):64-8. doi: 10.14712/fb2012058020064. PMID 22578956
- [Result] Fotouhi N, Ardalan M, Jabbarpour Bonyadi M, Abdolmohammadi R, Kamalifar A, Nasri H, Einollahi B. R229Q polymorphism of NPHS2 gene in patients with late-onset steroid-resistance nephrotic syndrome: a preliminary study. Iran J Kidney Dis. 2013 Sep;7(5):399-403. PMID 24072153
- [Result] Joshi S, Andersen R, Jespersen B, Rittig S. Genetics of steroid-resistant nephrotic syndrome: a review of mutation spectrum and suggested approach for genetic testing. Acta Paediatr. 2013 Sep;102(9):844-56. doi: 10.1111/apa.12317. Epub 2013 Jul 10. PMID 23772861